CLINICAL TRIAL: NCT01157923
Title: Evaluation of Automated Insulin Pump Settings Using the MD-Logic Pump Advisor-Adults Sub Study
Brief Title: MD Logic Pump Advisor- Adults Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rmc005816ctil
Record Dates: First submitted 2010-06-27; First posted 2010-07-07 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Type 1 Diabetes; Insulin Pump Therapy
Keywords: Type 1 diabetes; Insulin Pump Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervantion group (Experimental): Insulin pump settings (i.e., basal plan, correction factor, carbohydrate ration and insulin activity time) will be adjusted using the MD-Logic Pump Advisor.
  Interventions: Device: MD Logic Pump Advisor
- control group (No Intervention): Regular treatment, No change will be made in the insulin pump setting during the study(unless there is a medical need or any safety concern).

INTERVENTIONS:
Device: MD Logic Pump Advisor — Insulin pump settings (i.e., basal plan, correction factor, carbohydrate ration and insulin activity time) will be adjusted using the MD-Logic Pump Advisor
  Arms: intervantion group

SUMMARY:
Prospective, randomized, controlled, 30-78 days trial comparing MD-Logic pump algorithm to the standard of care of patients with type 1 diabetes.

The objective of this feasibility study is to evaluate the efficacy and safety of automated determined Insulin pump settings (i.e., basal plan, correction factor, carbohydrate ration and insulin activity time) using the MD-Logic Pump Advisor in individuals with type 1 diabetes.The study will be consisted from two segments:(I)pilot study, 30-78 days trial evaluating the MD-Logic pump advisor and (II)randomized controlled 30-78 days trial comparing MD-Logic pump algorithm to the standard of care.In segment 1, the pilot study, the aim is to enroll 15-30 subjects without control group. In segment 2, the randomized controlled segment, the aim is to enroll 92 subjects, but enrolling up to 105 eligible subjects to allow for dropouts.

The randomized controled study segment will be initiated after the pilot segment.Each segment of the study will consist of 6 clinic visits taking place at intervals of 1-3 weeks, sum of 30-78 days study duration for each segment. Before each clinic visit, subjects will wear continuous glucose sensors for 6 days; the intervention group will have up to 4 iterations (e.g the pump setting will be reviewed and adjusted up to 4 times during the study period according to the MD-Logic Pump Advisor).For the control group (at segment 2 only), insulin pump settings will not be changed during the study period (patient's usual standard of care).

DETAILED DESCRIPTION:
the MD-Logic Pump Advisor was design by the Diabetes Technology Center, the Institute of Endocrinology and Diabetes, National Center for Childhood Diabetes, Schneider Children's Medical Center of Israel. The MD-Logic Pump Advisor learns and adapts the patient's insulin pump settings in order to optimize glucose control. The MD-Logic Pump Advisor needs, as input, sensor readings, insulin delivery and recording of the meals during home care. During collection of the data, the patients are asked to continue their daily routine (no need for special consideration).

The present study was designed to test the automatic algorithm that will evaluate and change, when necessary, the patient's insulin pump settings based on prior sensor reading, insulin delivery, and meals data that was collected while the patient is under his regular treatment at home.

The objective of this feasibility study is to evaluate the efficacy and safety of automated determined Insulin pump settings (i.e., basal plan, correction factor, carbohydrate ration and insulin activity time) using the MD-Logic Pump Advisor in individuals with type 1 diabetes.

The study will be consisted from two segments:(I)pilot study, 30-78 days trial evaluating the MD-Logic pump advisor and (II)randomized controlled 30-78 days trial comparing MD-Logic pump algorithm to the standard of care.In segment 1, the pilot study, the aim is to enroll 15-30 subjects without control group. In segment 2, the randomized controlled segment, the aim is to enroll 92 subjects, but enrolling up to 105 eligible subjects to allow for dropouts.

The randomized controled study segment will be initiated after the pilot segment.Each segment of the study will consist of 6 clinic visits taking place at intervals of 1-3 weeks, sum of 30-78 days study duration for each segment. Before each clinic visit, subjects will wear continuous glucose sensors for 6 days; the intervention group will have up to 4 iterations (e.g the pump setting will be reviewed and adjusted up to 4 times during the study period according to the MD-Logic Pump Advisor).For the control group (at segment 2 only), insulin pump settings will not be changed during the study period (patient's usual standard of care).

Endpoints:

* Primary endpoint Increase in time spent in the normal range, defined as sensor glucose level within 70 to 180 mg/dl
* Secondary endpoints Reduced time spent above 180 mg/dl, reduced time spent below 70 mg/dl, reduced number of hypoglycemic events below 63 mg/dl, reduced glucose variability, quality of life measurements and subject treatment satisfaction.

Inclusion Criteria:

* Subject with Type 1 diabetes (>1yr since diagnosis)
* Medtronic ( MiniMed Paradigm 522, 512 , 722 or 712) insulin infusion pump CSII (continuous subcutaneous insulin infusion) therapy for at least 3 months
* Age ≥ 18 years
* HbA1c at inclusion ≥ 6.0%
* No concomitant diseases that influence metabolic control
* No current use of CGM
* Subjects do not participate in any other interventional study

ELIGIBILITY:
Inclusion Criteria:

1. Subject with Type 1 diabetes (>1yr since diagnosis)
2. Medtronic( MiniMed Paradigm 522, 512 , 722 or 712) insulin infusion pump CSII therapy for at least 3 months
3. Age ≥ 18 years
4. HbA1c at inclusion ≥ 6.0%
5. No concomitant diseases that influence metabolic control
6. No current use of CGM
7. Subjects do not participate in any other interventional study

Exclusion Criteria:

1. Known or suspected allergy to trial products.
2. Any significant diseases or conditions including psychiatric disorders and substance abuse that, in the opinion of the investigator, is likely to affect the subject's ability to complete the study, or compromise patient safety
3. Subject is currently using CGM device
4. Diabetic ketoacidosis in the past 3 months.
5. Severe hypoglycemia resulting in seizure or loss of consciousness in the month prior to enrollment.
6. Current use of oral glucocorticoids or other medications, which in the judgment of the investigator would be a contraindication to participation in the study.
7. Subject is participating in another drug or device study that could affect glucose measurements or glucose management.
8. Female subject who is pregnant or planning to become pregnant within the planned study duration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Time spent in the normal range | during each 6 days iteration
  increase in the time spent in the normal range, defined as sensor glucose level within 70-180 mg/dl

SECONDARY OUTCOMES:
number of iterations required to achieve the maximal meaningful improvement in the primary outcome | Day 78
  number of iterations required to achieve the maximal meaningful improvement in the primary outcome
time spent above 180 mg/dl | during each 6 days iteration
  time spent above 180 mg/dl
time spent below 70 mg/dl | during each 6 days iteration
  time spent below 70 mg/dl
Number of Hypoglycemic events below 63 mg/dl | during each 6 days iteration
  Number of Hypoglycemic events below 63 mg/dl
Adverse event | during each 6 days iteration
  Adverse event
glucose variability- area under the curve | during each 6 days iteration
  glucose variability measured as area under the curve (the area between the measured blood glucose and the glucose level of 180 mg/dl) and area above the curve (the area between the measured blood glucose and the glucose level of 70 mg/dl
Quality of Life Questionaires | At the end of the study- day 30 -78
  Quality of Life Questionaires
Number of MDLAP-recommendations that were rejected by the physician | during each 6 days iteration
  Number of MDLAP-recommendations that were rejected by the physician
Number and type of changes in any pump setting per iteration | during each 6 days iteration
  Number and type of changes in any pump setting per iteration

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, Prof, Principal Investigator — Schenider Children's Medical
Locations (2):
- Schneider Children's Medical center, Petaach-Tikva, Israel
- University Children's Hospital, Ljubljana, Slovenia